CLINICAL TRIAL: NCT07383909
Title: Evaluation of the Organ-Protective Effects of Remote Ischemic Preconditioning in Patients Undergoing Surgery for Acute Type A Aortic Dissection: A Multicenter, Prospective, Double-Blind, Randomized Controlled Trial
Brief Title: Remote Ischemic Preconditioning for Aute Type A Aortic Dissection Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, Chief, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A202601
Record Dates: First submitted 2025-12-08; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Aortic Dissection Type A
Keywords: Remote Ischaemic Conditioning; ischemia reperfusion injury; emergency surgery; major adverse outcomes
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC Intervention Group (Experimental): Participants randomized to this group will receive remote ischemic preconditioning (RIPC). After induction of general anesthesia, RIPC will be applied to the upper arm and thigh on the non-arterial cannulation side. The procedure consists of four alternating ischemia-reperfusion cycles, each cycle comprising 5 minutes of cuff inflation (at 200 mmHg, or systolic blood pressure +15 mmHg if systolic blood pressure exceeds 185 mmHg), followed by 5 minutes of cuff deflation for reperfusion. The inflation process alternates, starting with the upper arm. The thigh cuff inflation will begin only after the first upper arm inflation cycle is completed, and this process will repeat in alternating cycles.
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- Control Group (Sham Comparator): Participants randomized to this group will receive a sham RIPC procedure. The same cuff placement and timing as the experimental group are used, but the cuff is inflated to only 20 mmHg for 5 minutes followed by 5 minutes of deflation, simulating the RIPC procedure without inducing ischemia.
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — This intervention is a non-invasive organ protection procedure. After induction of general anesthesia, 4 cycles of remote ischemic preconditioning (RIPC) are applied to the upper arm and thigh on the non-arterial cannulation side. Each cycle consists of 5 minutes of cuff inflation (at 200 mmHg, or systolic blood pressure +15 mmHg if systolic blood pressure exceeds 185 mmHg) to induce ischemia, followed by 5 minutes of cuff deflation for reperfusion. To ensure safety, the cuff inflation cycles alternate between the upper arm and thigh. The procedure aims to activate endogenous protective mechanisms, enhancing the tolerance of vital organs to subsequent ischemic injury during surgery.

SUMMARY:
The goal of this clinical trial is to learn if a technique called remote ischemic preconditioning (RIPC) helps protect organs during emergency surgery for acute type A aortic dissection (ATAAD). The main questions it aims to answer are:

Does RIPC reduce the risk of major complications after surgery, such as heart, brain, or kidney problems?

Is RIPC safe to use during emergency ATAAD surgery?

Researchers will compare the RIPC group to a control group (who will receive a placebo) to see if RIPC can reduce complications after surgery.

Participants will:

Receive either RIPC or a sham intervention during their surgery.

Be monitored for up to 30 days after surgery for complications.

Have follow-up visits at 3 months, 1 year, and then yearly for up to 5 years to track their recovery.

DETAILED DESCRIPTION:
Study Design and Rationale

This study is a multicenter, prospective, double-blind, randomized, sham-controlled clinical trial designed to evaluate the organ-protective efficacy and safety of remote ischemic preconditioning (RIPC) in patients undergoing emergency surgery for acute type A aortic dissection (ATAAD).

Primary Objective

The primary objective of this study is to determine whether RIPC reduces the incidence of the primary composite endpoint of major adverse outcomes occurring from the time of surgery until hospital discharge (or up to 30 days postoperatively if hospitalization exceeds 30 days). This composite endpoint includes perioperative all-cause mortality and severe complications requiring invasive intervention or resulting in organ failure.

Key Interventions and Methodology Intervention Group

After induction of general anesthesia, patients in the intervention group receive the RIPC procedure. On the non-arterial cannulation side, alternating RIPC cycles are applied to both the upper arm and thigh, for a total of four cycles. The protocol begins with the upper arm cuff.

Each cycle consists of 5 minutes of cuff inflation (baseline pressure of 200 mm Hg; or at least 15 mm Hg above systolic pressure if systolic pressure exceeds 185 mm Hg), followed by 5 minutes of cuff deflation to allow reperfusion. The first cycle of the thigh cuff is initiated after completion of the first inflation cycle of the upper arm cuff.

Control Group

Patients in the control group undergo a sham procedure identical in timing and application sites to the RIPC intervention. However, the cuff is inflated to a low, non-ischemic pressure of 20 mm Hg for 5 minutes, followed by 5 minutes of deflation in each cycle.

Blinding

This study employs a double-blind design. Study participants, surgical teams, postoperative care providers, outcome assessors, and data analysts/statisticians are all blinded to treatment allocation. Only an independent researcher, who does not participate in subsequent patient assessment or data collection, is unblinded in order to perform the assigned intervention.

Standardization

All surgical procedures and perioperative care are conducted in accordance with standardized protocols at each participating center.

Study Endpoints Primary Endpoint

The incidence of the primary composite endpoint of major adverse outcomes from surgery until hospital discharge (or up to 30 days postoperatively).

Secondary Endpoints

Secondary endpoints include the incidence of each individual component of the primary composite endpoint at 30 days, 90 days, and 12 months postoperatively; the maximum SOFA-2 score within the first 3 postoperative days; surgery- and cardiopulmonary bypass-related times; duration of mechanical ventilation; lengths of intensive care unit (ICU) and hospital stay; postoperative all-cause mortality; and the rate of unplanned rehospitalization.

Quality Assurance and Data Management Site Selection and Training

Participating centers are required to have substantial experience in emergency ATAAD surgery. All investigators undergo centralized training on the study protocol and Standard Operating Procedures (SOPs), with a focus on the standardized RIPC procedure and data collection.

Clinical Monitoring

Clinical Research Associates (CRAs) conduct periodic on-site monitoring visits to ensure adherence to the study protocol and to verify consistency between data entered in the electronic Case Report Forms (eCRFs) and source documents.

Statistical Analysis

The primary analysis will be conducted in the intention-to-treat (ITT) population. Continuous variables will be compared using appropriate parametric or non-parametric tests, and categorical variables will be compared using the chi-square test or Fisher's exact test, as appropriate.

Sample Size Justification

Based on previously reported literature indicating an incidence of major adverse outcomes of approximately 25.8% after ATAAD surgery, and assuming an anticipated relative risk reduction of 26.5% with RIPC, sample size calculations using a two-sided alpha level of 0.05 and 80% statistical power determined that 589 evaluable patients are required per group. Allowing for an estimated dropout rate of 10%, the final target enrollment for this study is 1,296 patients.

Interim Analysis and Data Safety Monitoring

An independent Data and Safety Monitoring Board (DSMB) will oversee participant safety throughout the study and periodically review aggregated safety data.

A pre-specified blinded sample size re-estimation will be performed when approximately 600 participants have completed assessment of the primary endpoint. This analysis will be based on the pooled event rate and observed dropout rate only, without unblinding treatment allocation or conducting between-group efficacy comparisons. Therefore, the interim analysis will not affect the overall type I error rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, with no restriction on sex;
2. Diagnosis of acute Type A aortic dissection requiring emergency surgery (symptom onset <14 days);
3. Ability to understand the study objectives, voluntary provision of written informed consent by the patient or a legally authorized representative, and willingness to comply with follow-up.

Exclusion Criteria:

1. Traumatic or iatrogenic aortic dissection;
2. Previous open cardiac or thoracic aortic surgery;
3. Severe preoperative dysfunction of vital organs, such as persistent deep coma, abdominal compartment syndrome, or circulatory failure;
4. Severe comorbidities, including myocardial infarction within the past 7 days, stroke within the past 2 months; end-stage renal disease (eGFR <30 ml/min/1.73 m²); end-stage liver disease (total bilirubin >342 μmol/L or INR >2.0);
5. Evidence of ischemia in the limb planned for intervention, such as decreased skin temperature, pain, pallor, with or without sensory disturbance, paralysis, or diminished/absent pulses; or severe deformity or prior arteriovenous surgery at the intervention site;
6. Peripheral arterial disease involving the limbs, Raynaud phenomenon, active phlebitis, or a history of deep vein thrombosis of the lower extremities;
7. Current use of sulfonylurea oral hypoglycemic agents or nicorandil;
8. Life expectancy <1 year (e.g., advanced malignancy);
9. Participation in another clinical trial without having reached its primary endpoint;
10. Pregnancy or lactation; immunodeficiency (e.g., HIV positivity, history of organ transplantation); known bleeding disorders, coagulation abnormalities, or sickle cell anemia; active or uncontrolled infection;
11. Other severe physical or psychiatric disorders, or laboratory abnormalities, which in the investigator's judgment may increase risk or interfere with study outcomes, rendering the patient unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1296 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital major adverse outcomes | surgery to discharge or 30 days post-op
  A composite of major adverse outcomes (binary). Includes:
  Perioperative all-cause death;
  Severe post-op complications (Grade III/IV per IAASSG consensus), involving neurological, cardiovascular, respiratory, urinary, gastrointestinal, and other systems.

SECONDARY OUTCOMES:
Maximum SOFA-2 Score in First 3 Postoperative Days | From ICU admission (postoperatively) up to postoperative day 3
  The highest (peak) SOFA-2 score recorded during the first 3 days following surgery
Operative Time | During the surgical procedure
  Total duration of the surgical procedure from skin incision to skin closure, measured in minutes
Duration of Mechanical Ventilation | From end of surgery until extubation (assessed up to 30 days)
  Total time from the end of surgery until successful extubation, measured in hours. Re-intubation times are included if applicable
ICU Length of Stay | From ICU admission after surgery until ICU discharge (assessed up to 30 days)
  Total duration of stay in the Intensive Care Unit after surgery, measured in days
Hospital Length of Stay | From hospital admission for surgery until hospital discharge (assessed up to 30 days)
  Total duration of hospitalization after surgery, measured in days
All-cause mortality | 30 days, 90 days, 12 months, and every 12 months thereafter, up to 60 months
  All-cause mortality
Postoperative delirium | From the end of surgery until hospital discharge, assessed up to 30 days postoperatively
  Incidence of postoperative delirium
Unplanned readmission | 30 days, 90 days, 12 months, and every 12 months thereafter, up to 60 months
  The proportion of patients readmitted to the hospital within the follow-up period due to causes related to the original acute type A aortic dissection or its surgical treatment, excluding planned readmissions
Incidence of any individual component of the primary composite endpoint at 30 days, 90 days, and 12 months postoperatively | 30 days, 90 days, and 12 months postoperatively
  Incidence of each individual adverse event (including death, stroke, renal failure, reoperation, etc.) that constitutes the primary composite endpoint of Major Adverse Outcomes (MAO) at 30 days, 90 days, and 12 months after surgery.
Troponin I | Within postoperative day 3
  To observe changes in troponin I
Serum Creatinine | Within postoperative day 3
  To observe changes in serum creatinine

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Xiamen Cardiovascular Hospital, Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: No